CLINICAL TRIAL: NCT01091142
Title: Single-Ascending-Dose Safety and Tolerability Study of NP001 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Single-Ascending-Dose Safety/Tolerability of NP001 in Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuraltus Pharmaceuticals, Inc. (Industry)
Responsible Party: Nancy E. Isaac/VP Regulatory Affairs, Neuraltus Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NP001 Single Dose - ALS
Record Dates: First submitted 2010-03-19; First posted 2010-03-23 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NP001 (Experimental)
  Interventions: Drug: NP001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NP001 — Cohort 1: 0.3 mg/kg NP001(6:2 active:placebo) Cohort 2: 1.1 mg/kg NP001(6:2 active:placebo) Cohort 3: 2.1 mg/kg NP001(6:2 active:placebo) Cohort 4: 4.3 mg/kg NP001(6:2 active:placebo)
  Arms: NP001
Drug: Placebo — Cohort 1: placebo Cohort 2: placebo Cohort 3: placebo Cohort 4: placebo
  Arms: Placebo

SUMMARY:
Primary objectives: To assess the safety and tolerability of ascending doses of NP001 compared to placebo in subjects with ALS.

Secondary objective: To explore the effects of NP001 on biomarkers potentially relevant to ALS.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled single ascending dose safety and tolerability study. Approximately 32-56 subjects with clinical diagnosis of ALS according to modified El Escorial criteria are planned to receive a single dose of study drug, NP001.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 21 years - 75 years
* Subjects must be in generally sound health as appropriate for their ALS diagnosis.
* Subjects must have a clinical diagnosis of laboratory-supported probable or definite ALS, according to modified El Escorial criteria.
* Subjects receiving riluzole must be on a stable dose for at least 30 days prior to enrollment.
* Women of childbearing age must be non-lactating and surgically sterile or using an effective method of birth control and have a negative pregnancy test prior to dosing with study medication.
* Subjects must understand the study and be willing to adhere to protocol requirements as evidenced by provision of written informed consent.
* Subject must be willing and able to give signed informed consent that has been approved by the Institutional Review Board (IRB).
* Subjects must be willing to have an intravenous infusion.
* Subjects must have suitable veins for IV access as determined by examination.

Exclusion Criteria:

* Subjects should not require nor are expected to require life sustaining interventions for the next six months or longer. (e.g. invasive ventilation).
* Subjects must not have:

  * presence of a tracheotomy or invasive ventilation. Nocturnal non-invasive ventilation system (e.g. C-PAP) is allowed.
  * a diagnosis of neurologic disease known to mimic the muscle atrophy or weakness seen in ALS including MS, muscular dystrophy, spinal stenosis, peripheral neuropathy, inherited neuropathies or neuromuscular diseases, foramen magnum or brainstem tumor, or toxic conditions.
  * an active pulmonary disease under treatment including uncontrolled asthma, chronic obstructive pulmonary disease (pneumonia, bronchitis, etc.), pulmonary fibrosis, pulmonary infection in the last 2 months, or history of aspiration that may expose the subject to increased risk by participating in this trial as determined by the Investigator.
  * a history of unstable medical illness in the 3 months prior to screening including any emergent hospitalizations.
  * renal disease based on screening estimated creatinine clearance (eCcr) < 50 mL/minute (Cockcroft Gault estimate using ideal body weight) where:
  * evidence of elevated alanine aminotransferase greater than 3 times the upper limit of normal.
  * evidence of anemia, thrombocytopenia, or neutropenia (screening hematocrit <33%, platelet count < lower limit of normal for the site laboratory, or neutrophil count less than 1,500/mm3).
  * any condition that requires periodic red blood cell transfusions, erythropoietin or any blood dyscrasias undergoing active treatment in the past year.
  * clinical laboratory parameters that are clinically significant in the opinion of the Investigator.
  * systolic blood pressure in excess of 160 mmHg nor less than 100 mmHG or a diastolic blood pressure above 98 mmHg.
  * a history of G6PD deficiency (Glucose-6-phosphate dehydrogenase deficiency) determined by subject report.
  * a current history of hepatitis or HIV determined by subject report.
* Subjects must not be using systemic immunosuppressants including steroids and chemotherapeutic agents. Inhaled steroids, eye drops and local topical use are permitted with concurrence of Medical Monitor.
* Subjects must not have a hematologic disorder such as autoimmune anemia, or hemolytic anemia of any type including paroxysmal nocturnal hemoglobinuria or myoglobinuria.
* Subjects must not have a history of unexplained jaundice determined by subject report.
* Subjects must not have received IV Immunoglobulin (IG) within 30 days of the planned initial dose of study drug.
* Subjects must not be participating in another drug study or have participated in a drug study within the last 30 days prior to enrollment. Observational trials with no intervention are acceptable provided permission for the other study Sponsor is obtained in writing.
* Subjects must not have any other condition which in the Investigator's opinion would put the subject at risk by participating in this study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NP001 compared to placebo in subjects with ALS | 6 mo.

SECONDARY OUTCOMES:
To explore the effects of NP001 on biomarkers potentially relevant to ALS | 6 mo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Miller, MD, Principal Investigator — Forbes Norris ALS Treatment and Research, California Pacific Medical Center
Locations (3):
- United States (3):
  - California Pacific Medical Center, San Francisco, California
  - University of Kansas Medical Center - Landon Center on Aging, Kansas City, Kansas
  - Department of Neurology; University of Kentucky Medical Center, Lexington, Kentucky